CLINICAL TRIAL: NCT00786500
Title: Anti-diabetic Effect of Gynostemma Pentaphyllum Tea in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: Karolinska Institutet (Other); Swedish International Development Cooperation Agency (SIDA) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Diabetes II; Study 1
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2008-11

CONDITIONS: Type 2 Diabetes
Keywords: Herbal medicine; Type 2 diabetes; Insulin sensitivity; Insulin secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gynostemma pentaphyllum tea (Active Comparator)
  Interventions: Dietary Supplement: Gynostemma pentaphyllum tea
- Placebo tea (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo tea

INTERVENTIONS:
Dietary Supplement: Gynostemma pentaphyllum tea — 3 grams twice daily, orally
  Arms: Gynostemma pentaphyllum tea
Dietary Supplement: Placebo tea — 3 grams twice daily, orally
  Arms: Placebo tea

SUMMARY:
The aim of the present study was to investigate the long-term effects on blood glucose concentrations and possible adverse effects of an extract of Gynostemma pentaphyllum (GP). This is a plant growing in the mountain regions of Northern Vietnam and previously being used in traditional medicine. The GP extract, or placebo, was randomized to newly diagnosed patients with type 2 diabetes and administered as a "tea", 3 g two times daily during 12 weeks. All patients received instructions regarding diet and physical exercise. Oral glucose tolerance tests were performed at baseline and then every 4 weeks, and blood tests were taken with the purpose to monitor lipids, kidney and liver function, body weight and blood pressure.

DETAILED DESCRIPTION:
In Vietnam, herbal extracts have been used as a long-standing tradition to treat diabetic patients, but effects of these extracts have not been studied adequately. Based on previous results in experimental animals, we have selected the plant Gynostemma pentaphyllum (GP), which grows in the mountain region of Northern Vietnam. GP extract had a hypoglycemic effect on mice and rats, and was shown to contain a substance, phanoside, which stimulates insulin secretion. In addition, GP has been shown to reduce both hyperglycemia and hyperlipidemia in diabetic Zucker fatty rats.

The present study aimed at investigate effects of GP extract, administered as a "tea", and compared with placebo in a randomized, double-blind trial in drug-naive patients with newly diagnosed type 2 diabetes. All patients also received instructions about diet and physical exercise. In addition to monitoring effects on plasma glucose regulation, we also studied possible effects on plasma lipids, kidney and liver function as well as body weight and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, drug-naive patients with type 2 diabetes
* Fasting plasma glucose (FPG) 7.0-14.0 mmol/l
* HbA1c > 6%

Exclusion Criteria:

* Type 1 diabetes
* Liver failure
* Kidney Failure

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose | 12 weeks
HbA1c (glycosylated hemoglobin) | 12 weeks

SECONDARY OUTCOMES:
Liver enzymes (ALT, AST) | 12 weeks
Kidney function (S-creatinine, S-BUN) | 12 weeks
Plasma lipids (TG, Cholesterol, HDL-, LDL-) | 12 weeks
Blood pressure | 12 weeks
Body weight (BMI, hip-waist ratio) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claes Goran Ostenson, MD, PhD, Study Director — Karolinska Institutet
Locations (1):
- National Institute of Gerontology, HMU, Hanoi, Vietnam

REFERENCES:
- [Background] Hoa NK, Norberg A, Sillard R, Van Phan D, Thuan ND, Dzung DT, Jornvall H, Ostenson CG. The possible mechanisms by which phanoside stimulates insulin secretion from rat islets. J Endocrinol. 2007 Feb;192(2):389-94. doi: 10.1677/joe.1.06948. PMID 17283239
- [Background] Norberg A, Hoa NK, Liepinsh E, Van Phan D, Thuan ND, Jornvall H, Sillard R, Ostenson CG. A novel insulin-releasing substance, phanoside, from the plant Gynostemma pentaphyllum. J Biol Chem. 2004 Oct 1;279(40):41361-7. doi: 10.1074/jbc.M403435200. Epub 2004 Jun 25. PMID 15220351
- See also: Publication on the study — http://www.ncbi.nlm.nih.gov/pubmed/20213586